CLINICAL TRIAL: NCT02420717
Title: A Phase I-II Study of the Combination of Ruxolitinib or Dasatinib With Chemotherapy in Patients With Philadelphia Chromosome (Ph)-Like Acute Lymphoblastic Leukemia (ALL)
Brief Title: Ruxolitinib Phosphate or Dasatinib With Chemotherapy in Treating Patients With Relapsed or Refractory Philadelphia Chromosome-Like Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed early due to low accrual and lack of response.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0521; NCI-2015-00779 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0521 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Results first posted 2022-05-02 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Recurrent B Acute Lymphoblastic Leukemia; Recurrent Ph-Like Acute Lymphoblastic Leukemia; Refractory B Acute Lymphoblastic Leukemia; Refractory Ph-Like Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Cyclophosphamide; Cytarabine; Dasatinib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; ruxolitinib; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (ruxolitinib phosphate) (Experimental): Patients receive ruxolitinib phosphate PO BID. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin; Other: Laboratory Biomarker Analysis; Drug: Leucovorin; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Prednisone; Biological: Rituximab; Drug: Ruxolitinib Phosphate; Drug: Vincristine
- Cohort B (dasatinib) (Experimental): Patients receive dasatinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dasatinib; Drug: Dexamethasone; Drug: Doxorubicin; Other: Laboratory Biomarker Analysis; Drug: Leucovorin; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine
- Phase 1 (Experimental): Patients Receive ruxolitinib Phosphate PO BID. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin; Other: Laboratory Biomarker Analysis; Drug: Leucovorin; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Prednisone; Biological: Rituximab; Drug: Ruxolitinib Phosphate; Drug: Vincristine

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
  Arms: Cohort B (dasatinib)
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin — Given IV or PO
  Other Names: Folinic acid
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IV and PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi
  Arms: Cohort A (ruxolitinib phosphate); Phase 1
Drug: Vincristine — Given IV
  Other Names: Leurocristine; VCR; Vincrystine

SUMMARY:
This phase II trial studies the side effects and best dose of ruxolitinib phosphate and how well it works compared to dasatinib when given with chemotherapy in treating patients with Philadelphia chromosome-like acute lymphoblastic leukemia that has come back (relapsed) or has not responded to treatment (refractory). Ruxolitinib phosphate and dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving ruxolitinib phosphate or dasatinib with chemotherapy works better in treating patients with previously treated acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and maximal tolerated dose (MTD) of ruxolitinib phosphate (ruxolitinib) in combination with chemotherapy in patients with Philadelphia chromosome (Ph)-like acute lymphoblastic leukemia (ALL). (Phase I, ruxolitinib cohort only) II. To determine the response rate (complete response [CR]/CR with incomplete marrow recovery [CRi]) of ruxolitinib or dasatinib in combination with chemotherapy in patients with Ph-like ALL. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the response rate (CR/CRi) of ruxolitinib in combination with chemotherapy in patients with Ph-like ALL. (Phase I, ruxolitinib cohort only) II. To determine the duration of response, disease-free survival and overall survival of ruxolitinib in combination with chemotherapy in patients with Ph-like ALL. (Phase I, ruxolitinib cohort only) III. To determine the safety and toxicity profile of ruxolitinib or dasatinib in combination with chemotherapy in patients with Ph-like ALL. (Phase II) IV. To determine the duration of response, disease-free survival and overall survival of ruxolitinib or dasatinib in combination with chemotherapy in patients with Ph-like ALL. (Phase II)

OUTLINE: This is a phase I, dose escalation study of ruxolitinib followed by a phase II study. Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients receive ruxolitinib phosphate orally (PO) twice daily (BID). Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

COHORT B: Patients receive dasatinib PO once daily (QD). Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

INTENSIVE CHEMOTHERAPY: After cycle 1, patients not achieving a response also receive cyclophosphamide intravenously (IV) over 3 hours BID on days 1-3, doxorubicin IV over 24-48 hours on day 4, vincristine IV over 30 minutes on days 4 and 11, and dexamethasone PO QD or IV over 30 minutes on days 1-4 and 11-14 of cycles 1, 3, 5, and 7. Patients receive methotrexate IV over 24 hours on day 1, leucovorin IV over 1 hour or PO every 6 hours on days 2-5, cytarabine IV over 2 hours BID on days on days 2 and 3 of cycles 2, 4, 6, and 8. At the discretion of the treating physician, patients may also receive rituximab IV over several hours on days 1 and 11 of cycles 1 and 3 and on days 1 and 8 of cycles 2 and 4 only. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive mercaptopurine PO thrice daily (TID), methotrexate PO once a week, vincristine IV over 30 minutes on day 1, and prednisone PO on days 1-5. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously treated B-cell ALL (relapsed and/or refractory after prior therapy)
* Bone marrow involvement with >= 5% lymphoblasts
* Documented genetic lesion(s) known to confer susceptibility to inhibition by either ruxolitinib or dasatinib or cytokine receptor-like factor 2 (CRLF2) positivity by flow cytometry (for the ruxolitinib cohort)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin < 2.0 mg/dL
* Serum glutamate pyruvate transaminase (SGPT) or serum glutamic oxaloacetic transaminase (SGOT) < 3 x upper limit of normal (ULN)
* Creatinine < 2 mg/dL
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (beta-hCG) pregnancy test result within 14 days prior to the first dose of study drugs and must agree to use an effective contraception method during the study and for 30 days following the last dose of study drug; females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy; appropriate methods of birth control include the following: any 2 of the following methods used together: birth control implants, injections, or pills (except for progesterone only pills), intrauterine device (IUD), vasectomy, tubal ligation, barrier method (female or male condom with spermicide, cervical cap with spermicide, diaphragm with spermicide); male condom with spermicide and diaphragm; male condom with spermicide and cervical cap; unacceptable methods of birth control include using no birth control, withdrawal, rhythm method, vaginal sponge, any barrier method that does not use spermicide, progesterone only pills, and using male and female condoms at the same time
* Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 30 days following the last dose of study drug
* Patients or their legally authorized representative must provide written informed consent

Exclusion Criteria:

* Burkitt's leukemia or lymphoma, T-cell ALL or lymphoblastic lymphoma
* Patients having undergone prior allogeneic stem cell transplant within 3 months or having active graft versus host disease
* Patient is pregnant or breastfeeding
* Patients with uncontrolled active infections (fever >= 38 degrees Celsius [C], septic shock)
* Isolated extramedullary relapse (i.e. testicular, central nervous system)
* Current or chronic hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
* Concurrent chemotherapy (except intrathecal chemotherapy)
* Major surgery within 4 weeks prior to first study dose
* Systemic chemotherapy/radiotherapy/investigational therapy within 14 days (with the exception of hydroxyurea and steroids) prior to starting therapy; for patients receiving ALL maintenance with 6-mercaptopurine, methotrexate, vincristine, and steroids - these agents should be discontinued at least 48 hours prior to start of study drugs; for patients on oral targeted therapies (such as imatinib, dasatinib, ponatinib), - these agents should be discontinued at least 48 hours prior to start of study drugs
* Patients must have recovered from acute non hematologic toxicity (to =< grade 1) of all previous therapy prior to enrollment
* Known active central nervous system (CNS) leukemia, as defined by unequivocal morphologic evidence of lymphoblasts in the cerebrospinal fluid (CSF), use of CNS-directed local treatment for active disease within the prior 28 days, symptomatic CNS leukemia (i.e., cranial nerve palsies or other significant neurologic dysfunction) within 28 days; patients may have history of CNS leukemic involvement if definitively treated with prior therapy and no evidence of active disease (defined as >= 2 consecutive spinal fluid assessments with no evidence of disease) at the time of registration; prophylactic intrathecal chemotherapy is not a criterion for exclusion
* Patients with active heart disease (New York Heart Association [NYHA] class 3-4 as assessed by history and physical examination, unstable angina/stroke/myocardial infarction within the last 6 months)
* Patients with a cardiac ejection fraction (as measured by either multi-gated acquisition [MUGA] scan or echocardiogram) < 40%; (Note: patients who have had prior anthracycline exposure of > 250 mg/m^2 may be eligible after discussion with the principal investigator [PI])
* Second malignancy other than basal cell or squamous cell carcinoma of the skin or in situ carcinoma of the cervix or the breast, unless they are successfully treated with curative intent for more than 2 years before entering the study
* Malabsorption syndrome or other conditions that preclude enteral route of administration
* Patients requiring strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 2015 to March 2020
Pre-assignment Details: There were no participants enrolled in the phase II portion of this study, the study did not move on to phase II due to slow accrual and lack of response.
Groups:
- Phase I Ruxolitinib 15mg; Phase I Ruxolitinib 20mg; Phase I Ruxolitinib 25mg: Patients receive Ruxolitinib phosphate PO BID. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I Ruxolitinib 15mg | Phase I Ruxolitinib 20mg | Phase I Ruxolitinib 25mg
Started | 5 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 2 | 0 | 0
Not completed — Did not receive all study medication | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Ruxolitinib 15mg | Phase I Ruxolitinib 20mg | Phase I Ruxolitinib 25mg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 3 | 11
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 24 [18 to 58] | 21 [20 to 62] | 44 [28 to 60] | 24 [18 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 3
  Male | 3 | 2 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 3 | 3 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximal Tolerated Dose (MTD) of Ruxolitinib in Combination With Chemotherapy Defined as the Highest Dose Level at Which no More Than 1 Out of 6 Patients Experience a Dose Limiting Toxicity (Phase I)
Description: The method of Thall, Simon and Estey will be used for toxicity monitoring for this study. The severity of the toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 whenever possible. Safety data will be summarized by category, severity and frequency.
Time Frame: 42 days
Population: Two out of nine participants were not Analyzed for response because they did not receive all planned study medication.
Measure: Number; unit: Milligrams (mg)
Arm/Group | Phase I Ruxolitinib 15mg
Number analyzed (Participants) | 9
Milligrams (mg) | 25

2. Primary Outcome: Participants With Complete Response (Complete Response [CR]/CR With Incomplete Marrow Recovery [CRi]) (Phase II)
Description: Complete Response (CR) is disappearance of all clinical and/or radiologic evidence of disease, Neutrophil count ≥ 1.0 x 10^9/L, Platelet count ≥ 100 x 10^9/L, Normal bone marrow differential (≤ 5% blasts), No extra-medullary leukemia. Complete Remission with Incomplete Blood Count Recovery (CRi) is CR except for ANC < 1.0 x 10^9/L and/or platelets < 100 x 10^9/L.
Time Frame: 42 days
Population: Two out of five participants in the Ruxolitinib 15mg arm were not Analyzed for response because they did not receive all planned study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Ruxolitinib 15mg | Phase I Ruxolitinib 20mg | Phase I Ruxolitinib 25mg
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 1 | 0

3. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 4 years 7 months
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I Ruxolitinib 15mg | Phase I Ruxolitinib 20mg | Phase I Ruxolitinib 25mg
Number analyzed (Participants) | 3 | 3 | 3
Months | 4.8 [2.4 to 11.3] | 5.4 [1.4 to 16.3] | 38.5 [4.9 to 41.9]

4. Secondary Outcome: Progression-free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 4 years 7 months
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I Ruxolitinib 15mg | Phase I Ruxolitinib 20mg | Phase I Ruxolitinib 25mg
Number analyzed (Participants) | 3 | 3 | 3
Months | 2.3 [1.5 to 11.3] | 1.8 [1.3 to 5.4] | 1.9 [1.8 to 3.1]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Phase I Ruxolitinib 15mg | Phase I Ruxolitinib 20mg | Phase I Ruxolitinib 25mg
All-Cause Mortality (participants affected / at risk) | 2/5 | 1/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 3/3
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Ruxolitinib 15mg (N=5) | Phase I Ruxolitinib 20mg (N=3) | Phase I Ruxolitinib 25mg (N=3)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Blood Antidiuretic Hormone Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
General Disorders and Administration Site Conditions, Other (General disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Infection and Infestations - other (Infections and infestations) | 0 (0) | 2 (3) | 1 (1)
Lung Infection (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Ruxolitinib 15mg (N=5) | Phase I Ruxolitinib 20mg (N=3) | Phase I Ruxolitinib 25mg (N=3)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alkaline Phosphatase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Back Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Blood Bilirubin Increase (Investigations) | 2 (2) | 1 (1) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Creatinine Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Eye Disorders - Other (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Infections and Infestations Other (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Investigations (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nervous System Disorders (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pain Extremity (General disorders) | 1 (1) | 0 (0) | 0 (0)
Psychiatric Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and Urinary Disorders (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT02420717/Prot_SAP_000.pdf